CLINICAL TRIAL: NCT03170154
Title: Clinical Investigation of the Clareon® IOL
Brief Title: Clinical Investigation of the Clareon® Intraocular Lens (IOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILJ466-C001
Record Dates: First submitted 2017-05-26; First posted 2017-05-30 (Actual); Results first posted 2020-03-09 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Clareon IOL (Experimental): Clareon aspheric hydrophobic acrylic monofocal IOL implanted in one eye during routine small incision cataract surgery
  Interventions: Device: Clareon aspheric hydrophobic acrylic monofocal IOL

INTERVENTIONS:
Device: Clareon aspheric hydrophobic acrylic monofocal IOL — Ultraviolet-absorbing and blue light-filtering IOL composed of high refractive-index foldable and flexible acrylic material. IOLs are implantable medical devices intended for long term use over the lifetime of the cataract subject.

SUMMARY:
The objective of this study is to compare visual acuity and adverse event outcomes from the Clareon intraocular lens (IOL) to historical safety and performance endpoint (SPE) rates.

DETAILED DESCRIPTION:
Upon meeting eligibility criteria, subjects were implanted unilaterally (in one eye) with a Clareon IOL. Subjects attended 7 study visits over a period of approximately 13 months, including 1 preoperative screening visit (Visit 0), 1 operative visit (Visit 00), and 5 postoperative visits (Visits 1-5). Visit day calculations for Visits 1-5 were based off of the day of surgery (Visit 00). Primary endpoint data was collected at the final visit (Month 12). Some sites/subjects participated in a Rotational Stability sub-study. For the non-study eye, the investigator followed standard of care regarding the follow-up, surgery, and intraocular lens choice (as applicable). The non-study eye (fellow eye) was not implanted with the Clareon IOL.

ELIGIBILITY:
Key Inclusion Criteria:

* Planned routine cataract surgery in at least one eye;
* Calculated lens power within the available range;
* Willing and able to sign an informed consent statement;
* Clear intraocular media other than cataract.

Key Exclusion Criteria:

* Any disease or pathology, other than cataract, that is expected to reduce the potential postoperative best corrected distance visual acuity (BCDVA) to a level worse than 0.30 logMAR;
* Previous corneal surgery;
* Rubella or traumatic cataract;
* Ocular trauma, previous refractive surgery;
* Current or recent use of certain medications as specified in the protocol;
* Any other ocular or systemic condition that, in the opinion of the Investigator, should exclude the subject from the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Surgical, Study Director — Alcon Research, LLC
Locations (16):
- United States (16):
  - Alcon Investigative Site, Fresno, California
  - Alcon Investigative Site, Sacramento, California
  - Alcon Investigative Site, San Leandro, California
  - Alcon Investigative Site, Deerfield Beach, Florida
  - Alcon Investigative Site, Orland Park, Illinois
  - Alcon Investigative Site, Bloomfield Hills, Michigan
  - Alcon Investigative Site, Kansas City, Missouri
  - Alcon Investigative Site, New York, New York
  - Alcon Investigative Site, Poughkeepsie, New York
  - Alcon Investigative Site, Elizabeth City, North Carolina
  - Alcon Investigative Site, Southern Pines, North Carolina
  - Alcon Investigative Site, Florence, South Carolina
  - Alcon Investigative Site, Ladson, South Carolina
  - Alcon Investigative Site, Austin, Texas
  - Alcon Investigative Site, Nacogdoches, Texas
  - Alcon Investigative Site, Appleton, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 16 investigative sites located in the United States.
Pre-assignment Details: Of the 376 enrolled, 26 subjects did exit the study as screen failures. This reporting group (350) includes all subjects with attempted implantation with the IOL (successful or aborted after contact with the eye).
Groups:
- Clareon IOL: Clareon aspheric hydrophobic acrylic monofocal intraocular lens (IOL) implanted in one eye during routine small incision cataract surgery
Period: Overall Study
Arm/Group | Clareon IOL
Started | 350
Rotational Stability Sub-study | 141
Completed | 342
Not Completed | 8
Not completed — Lost to Follow-up | 4
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: All-Implanted (AAS): All subjects with successful IOL implantation
Arm/Group | Clareon IOL
Number analyzed (Participants) | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (6.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213
  Male | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 336
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 36
  White | 273
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 350

OUTCOME MEASURES:

1. Primary Outcome: Percentage of All-implanted Subjects Achieving Monocular Best Corrected Distance Visual Acuity (BCDVA) of 0.3 logMAR or Better at Month 12 Postoperative
Description: Visual acuity (VA) of the study eye was assessed with best refractive correction in place under photopic (well-lit) conditions at a distance of 4 meters using Early Treatment Diabetic Retinopathy Study (ETDRS) letter charts. As pre-specified in the protocol, the percentage of subjects with monocular BCDVA of 0.3 logMAR or better at Month 12 was compared to the historical safety and performance endpoint (SPE) rate reported in EN ISO 11979-7:2014. A higher percentage indicates good visual acuity outcomes with most subjects achieving 0.3 logMAR or better.
Time Frame: Month 12 (postoperative)
Population: All-Implanted Subjects (AAS): All subjects/eyes with successful IOL implantation and data at visit
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | Clareon IOL
Number analyzed (Participants) | 342
Number analyzed (eyes) | 342
percentage of subjects | 99.7 [98.38 to 99.99]
Statistical Analysis 1: Comparison: Clareon IOL; Test type: Other; 1-sided 95% Upper CL = 99.99 — Historical comparison to EN ISO 11979-7:2014: SPE rate of at least 92.5 for the AAS at 12 months

2. Primary Outcome: Percentage of Best-case Subjects Achieving Monocular BCDVA of 0.3 logMAR or Better at Month 12 Postoperative
Description: Visual acuity (VA) of the study eye was assessed with best refractive correction in place under photopic conditions at a distance of 4 meters using an Early Treatment Diabetic Retinopathy Study (ETDRS) letter charts. As pre-specified in the protocol, the percentage of subjects with monocular BCDVA of 0.3 logMAR or better at Month 12 was compared to the historical safety and performance endpoint (SPE) rate reported in EN ISO 11979-7:2014. A higher percentage indicates good visual acuity outcomes with most subjects achieving 0.3 logMAR or better.
Time Frame: Month 12 (postoperative)
Population: Best-Case Analysis Set (BAS): All subjects/eyes successfully implanted with the IOL that had at least 1 postoperative visit, no preoperative ocular pathology, no macular degeneration at any time, and no previous surgery for the correction of refractive errors, with data at visit.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Units Other Than Participants: eyes
Arm/Group | Clareon IOL
Number analyzed (Participants) | 326
Number analyzed (eyes) | 326
percentage of subjects | 99.7 [98.30 to 99.99]
Statistical Analysis 1: Comparison: Clareon IOL; Test type: Other; 1-sided 95% Upper CL = 99.98 — Historical comparison to EN ISO 11979-7:2014: SPE rate of at least 96.7 for the BAS at 12 months

3. Primary Outcome: Percentage of Subjects With Adverse Events (Ocular and Nonocular, Serious and Nonserious), Including Secondary Surgical Interventions (SSIs) - Study Eye
Description: Adverse events (AEs) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. No hypothesis testing was pre-specified in the protocol.
Time Frame: Day 0 (operative), up to Month 12 (postoperative)
Population: Safety Analysis Set (SAS): All subjects/study eyes with attempted implantation with the test article (successful or aborted after contact with the eye)
Measure: Number; unit: percentage of subjects
Groups:
- Pre-treatment: Events reported in this group occurred prior to attempted implantation with the test article and may include ocular events in the study eye, as well as overall systemic events.
- Clareon IOL - Ocular: Events reported in this group occurred after attempted implantation with the test article and include ocular events in the study eye.
- Systemic: Events reported in this group occurred after attempted implantation with the test article.
Arm/Group | Pre-treatment | Clareon IOL - Ocular | Systemic
Number analyzed (Participants) | 350 | 350 | 350
percentage of subjects
  Serious Adverse Events | 0 | 2.3 | 4.0
  Non-Serious Adverse Events | 1.4 | 27.1 | 15.1

4. Secondary Outcome: Mean Absolute IOL Rotation
Description: IOL rotation was defined as the difference between axis of IOL orientation on the day of surgery and Month 6. IOL rotation and measured with slit-lamp photography. No hypothesis testing was pre-specified in the protocol. A lower number indicates minimal IOL rotation at 6 months.
Time Frame: Day 0 (operative), Month 6 (postoperative)
Population: Rotation Analysis Set (RAS): All subjects/eyes with successful IOL implantation from the rotational subset of 6 clinical sites, with rotation data available at operative visit and Month 6 visit.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: eyes
Arm/Group | Clareon IOL
Number analyzed (Participants) | 124
Number analyzed (eyes) | 124
degrees | 2.2696 (3.87231)

5. Secondary Outcome: Mean Absolute IOL Misplacement
Description: IOL misplacement was defined as the difference between intended axis of placement and actual axis of IOL orientation on day of surgery. IOL misplacement was measured using slit lamp photography. No hypothesis testing was pre-specified in the protocol. A lower number indicates minimal IOL misplacement.
Time Frame: Day 0 (operative)
Population: RAS: All subjects/eyes with successful IOL implantation from the rotational subset of 6 clinical sites, with rotation data available at operative visit.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: eyes
Arm/Group | Clareon IOL
Number analyzed (Participants) | 131
Number analyzed (eyes) | 131
degrees | 5.1163 (4.90305)

6. Secondary Outcome: Mean Absolute IOL Misalignment
Description: IOL misalignment was defined as the summation of IOL misplacement and IOL rotation at Month 6. No hypothesis testing was pre-specified in the protocol. A lower number indicates minimal IOL misalignment at 6 months.
Time Frame: Day 0 (operative), Month 6 (postoperative)
Population: RAS, with rotation data available at operative visit and Month 6 visit
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: eyes
Arm/Group | Clareon IOL
Number analyzed (Participants) | 124
Number analyzed (eyes) | 124
degrees | 5.6762 (6.42510)

ADVERSE EVENTS:
Time Frame: Adverse events were collected pre-treatment (Day -30 to 0) up to Month 12 post-treatment/study exit. Adverse events (AEs) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator.
Description: This analysis population includes all subjects/eyes with attempted implantation with the test article (successful or aborted after contact with the eye). "At Risk" population of pre-treatment and systemic AEs is reported in units of subjects; ocular AE population is reported in units of eyes. For the non-study eye (fellow eye), the investigator followed standard of care regarding the follow-up, surgery, and IOL choice (as applicable). The non-study eye was not implanted with Clareon IOL.
Groups:
- Pre-treatment: Events reported in this group occurred prior to attempted implantation with the test article and may include ocular events in the study eye and non-study eye (fellow eye), as well as overall systemic events. The non-study eye was not implanted with Clareon IOL.
- Clareon IOL - Ocular (Study Eye): Events reported in this group occurred after attempted implantation with the test article and include ocular events in the study eye.
- Systemic and Ocular Non-Study (Non-Clareon) Eye: Events reported in this group occurred after attempted implantation with the test article and may include ocular events in the non-study eye (fellow eye), as well as overall systemic events. The non-study eye was not implanted with Clareon IOL.
Arm/Group | Pre-treatment | Clareon IOL - Ocular (Study Eye) | Systemic and Ocular Non-Study (Non-Clareon) Eye
All-Cause Mortality (participants affected / at risk) | 0/350 | 0/350 | 2/350
Serious Adverse Events (participants affected / at risk) | 0/350 | 8/350 | 18/350
Other Adverse Events (participants affected / at risk) | 6/350 | 19/350 | 127/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-treatment (N=350) | Clareon IOL - Ocular (Study Eye) (N=350) | Systemic and Ocular Non-Study (Non-Clareon) Eye (N=350)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cystoid macular oedema (Eye disorders) | 0 (0) | 3 (3) | 1 (1)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Punctate keratitis (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Retinal tear (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Corneal operation (Surgical and medical procedures) | 0 (0) | 1 (2) | 2 (2)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Ophthalmologic treatment (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Radical hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Retinal laser coagulation (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Retinopexy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Urostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Vitrectomy (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-treatment (N=350) | Clareon IOL - Ocular (Study Eye) (N=350) | Systemic and Ocular Non-Study (Non-Clareon) Eye (N=350)
Posterior capsule opacification (Eye disorders) | 0 (0) | 19 (19) | 18 (18)
Cataract operation (Surgical and medical procedures) | 6 (6) | 0 (0) | 117 (117) — Pre-planned cataract operations in the non-study eye (non-Clareon eye) (fellow eye) are recorded as adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT03170154/SAP_000.pdf
  • Study Protocol (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT03170154/Prot_001.pdf